CLINICAL TRIAL: NCT03641716
Title: Family Empowerment for Enhanced Development
Acronym: Project FEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Angela Caldwell, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO17070504; UL1TR001857 (NIH)
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Results first posted 2021-01-08 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Obesity, Childhood; Feeding Behavior
Keywords: early childhood, family, occupational therapy
MeSH Terms: conditions — Pediatric Obesity; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Repeated Measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mealtime PREP Intervention (Experimental): Parents of young children will receive 6 weekly sessions, each lasting approximately one-hour, in the home environment. An occupational therapy clinician will deliver the Mealtime PREP intervention to the family.
  Interventions: Behavioral: Mealtime PREP Intervention

INTERVENTIONS:
Behavioral: Mealtime PREP Intervention — Each session will include didactic elements and skills training along with skills practice and feedback. Parents will learn to build structured mealtime routines, manage child mealtime behavior, and incorporate exploration and play into routines.
  Other Names: Promoting Routines of Exploration and Play during Mealtime

SUMMARY:
This study evaluates the feasibility and preliminary effects of offering the Mealtime PREP intervention to low-income families with young children. All enrolled families will receive the Mealtime PREP intervention in the home to evaluate the effects on child nutrition.

DETAILED DESCRIPTION:
Children have not been spared from the obesity epidemic. There is a great need for innovative interventions to help families build healthy habits early in life for obesity prevention. Low-income preschoolers have a disproportionately high rate of childhood obesity, and their families face complex barriers to healthy behavior change. This proposed pilot study will examine the feasibility of delivering the Promoting Routines of Exploration and Play during Mealtime (Mealtime PREP) intervention in a sample of low-income families with young children (ages 2-5). Our parent-mediated intervention is designed to promote healthy dietary variety using routine family meals, positive reinforcement, social modeling, and food exploration and play. By harnessing the behavior change capacity of behavioral activation to alter daily mealtimes incrementally, parents are empowered to overcome barriers to healthy habit formation. Each family will participate in a six-week intervention that is delivered by occupational therapy clinicians in the home environment. Each session will last approximately one hour and include individualized parent-training and a parent-led mealtime with direct feedback from the clinician. We planned to screen up to 100 potential parent and child participants, with a plan to deliver intervention to 20 child participants.

ELIGIBILITY:
Inclusion Criteria:

Child:

* within age range 2-5 years
* reside in a low-income household (as specified by income within the range to qualify for Special Supplemental Nutrition Program for Women, Infants, and Children.

Parent:

* >18 years old
* ability to read and speak in English
* willing to participate in 6 home-based intervention sessions

Exclusion Criteria:

* None

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela R Caldwell, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between February and June of 2019 using research registry (Pitt + Me) and in the community at WIC (Supplemental Nutrition for Women, Infants and Children) program sites.
Groups:
- Mealtime PREP Intervention: Parents of young children will receive 6 weekly sessions, each lasting approximately one-hour, in the home environment. An occupational therapy clinician will deliver the Mealtime PREP (Promoting Routines of Exploration and Play) intervention to the family.
  Mealtime PREP Intervention: Each session will include didactic elements and skills training along with skills practice and feedback. Parents will learn to build structured mealtime routines, manage child mealtime behavior, and incorporate exploration and play into routines.
Period: Overall Study
Arm/Group | Mealtime PREP Intervention
Started | 20
Completed | 15
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Mealtime PREP Intervention
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 43.76 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 5
  More than one race | 4
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20
3-Day Food Diary [Mean (Standard Deviation); unit: number of unique foods] — The 3-Day Food Diary is the preferred method of dietary assessment (intake and variety of food consumed) because of a balance between validity and burden. Includes all food consumed and approximate servings for 3 days. Servings of foods consumed from each food group will be tallied and compared to national daily recommendations. Population: We only received 3-Day Food Diaries back from 3 participants at baseline.
  number of unique foods
    number analyzed (Participants) | 3
    (all) | 19 (5)
Parenting Stress Index - Short Form [Mean (Standard Deviation); unit: units on a scale] — 36 item scale validated in a sample of low-income families with preschoolers to assess parental stress in three domains and overall. Raw scores are converted to percentiles for interpretation using this tool. For the total parenting stress score, and all three domain scores (Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child), higher percentiles are interpreted as higher stress (range =1-99%) with scores >90% indicating clinically significant levels of parenting stress. We are reporting the Total parenting stress score. Population: Missing data led to inability to score baseline PSIs for 8 participants
  units on a scale
    number analyzed (Participants) | 12
    (all) | 75.67 (30.16)
Nutrition Screening Tool for Every Preschooler [Mean (Standard Deviation); unit: units on a scale] — 17 item, validated screen for young children (1-5 years) that categorizes risk of nutritional problems into 3 categories (score range = 1 (minimum) - 68 (maximum); 1 - 20 = low risk, 21-25 = moderate risk, and 26+ = high risk). Higher scores indicate higher risk for nutritional problems (i.e. lower scores are better).
  units on a scale | 22.90 (8.94)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline 3-Day Food Diary (Dietary Variety) at 3 Months
Description: The 3-Day Food Diary is the preferred method of dietary assessment (intake and variety of food consumed) because of a balance between validity and burden. Includes all food consumed and approximate servings for 3 days. Servings of foods consumed from each food group will be tallied and compared to national daily recommendations. We calculated the number of unique foods consumed at baseline and the 3-month follow-up.
Time Frame: baseline and 3 months
Population: We only received completed 3-Day Food Diaries from three participants at both baseline and the 3-month follow-up time frame.
Measure: Mean (Standard Deviation); unit: number of unique foods
Arm/Group | Mealtime PREP Intervention
Number analyzed (Participants) | 3
number of unique foods | 3.66 (2.08)
Statistical Analysis 1: Comparison: Mealtime PREP Intervention; Test type: Other; Mean Difference (Net) = 3.67, Standard Deviation 2.08

2. Secondary Outcome: Change From Baseline Parenting-Stress Inventory, Short-Form (PSI-SF) to 3 Months
Description: 36 item scale validated in a sample of low-income families with preschoolers to assess parental stress in three domains and overall. Raw scores are converted to percentiles for interpretation using this tool. For the total parenting stress score, and all three domain scores (Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child), higher percentiles are interpreted as higher stress (range =1-99%) with scores >90% indicating clinically significant levels of parenting stress. We are reporting the Total parenting stress score.
Time Frame: Baseline, 3 months
Population: We experienced a significant amount of missing data for the first 8 participants completing this form, which led to an inability to calculate scores for baseline. Research procedures were adjusted, but only had complete data on 9 of 12 remaining participants at 3 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mealtime PREP Intervention
Number analyzed (Participants) | 9
score on a scale | 0.22 (25.04)
Statistical Analysis 1: Comparison: Mealtime PREP Intervention; Due to limited size of sub-sample, we calculated a Cohen's d effect size for raw total score on the PSI from baseline to the 3-month follow-up, with a 95% confidence interval; Test type: Other; Effect Size - Cohen's d = -.01, 95% CI 2-sided [-.66 to .65]

3. Secondary Outcome: Change From Baseline Nutrition Screening Tool for Every Preschooler (Nutritional Risk) at 3 Months
Description: 17 item, validated screen for young children (1-5 years) that categorizes risk of nutritional problems into 3 categories (score range = 1 (minimum) - 68 (maximum); 1 - 20 = low risk, 21-25 = moderate risk, and 26+ = high risk). Higher scores indicate higher risk for nutritional problems (i.e. lower scores are better).
Time Frame: baseline and 3 months
Population: 5 participants lost to follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mealtime PREP Intervention
Number analyzed (Participants) | 15
score on a scale | -2.80 (5.43)
Statistical Analysis 1: Comparison: Mealtime PREP Intervention; After examining the data to ensure it met the statistical assumptions (e.g. normality, no outliers), we ran a paired-sample pre-post t-test to examine the difference in scores from baseline to 3 months on the NutriSTEP (Screening Tool for Every Preschooler) assessment; Test type: Other; p < .01, t-test, 2 sided — a prior threshold for statistical significance set at p<.05; We ran a paired samples t-test with pre/post intervention data (from baseline and 3-month assessments)

ADVERSE EVENTS:
Time Frame: We collected data on adverse events during our intervention period (6 weeks)
Arm/Group | Mealtime PREP Intervention
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
This clinical trial is limited by small sample size and difficulty obtaining 3-Day Food Diaries (as participants had to mail these back in a pre-stamped and addressed envelope after completion). No inferences can be made regarding changes observed in the 3-Day food Diary due to this limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT03641716/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT03641716/ICF_001.pdf